CLINICAL TRIAL: NCT04245345
Title: Accelerometer Sensing for Micra AV Study
Acronym: AccelAV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AccelAV
Record Dates: First submitted 2020-01-21; First posted 2020-01-28 (Actual); Results first posted 2023-02-13 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: AV Block; AV Block Complete; 3rd Degree Heart Block; Complete Heart Block
Keywords: AV Synchrony; Micra AV; Micra; Transcatheter Pacing; Normal Sinus Node Function; Leadless Pacemaker
MeSH Terms: conditions — Atrioventricular Block

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Single-arm (Other): Subjects implanted with the Medtronic Micra AV device
  Interventions: Device: Accelerometer Sensing for Micra AV Study

INTERVENTIONS:
Device: Accelerometer Sensing for Micra AV Study — Characterize AV synchrony in subjects implanted with Micra AV device. The study will be conducted upon market approval of the Micra AV Transcatheter Pacing System.

SUMMARY:
The purpose of the AccelAV Study is to characterize chronic AV synchrony in subjects implanted with MicraTM AV device. This study will be conducted upon market approval of the MicraTM AV Transcatheter Pacing System.

DETAILED DESCRIPTION:
The Accel AV study is a prospective, single-arm, global, multi-center clinical study to characterize the chronic AV synchrony in subjects implanted with the market released Micra AV system. The study is planned to be conducted in the US and Hong Kong. Overall, the study is expected to be conducted at approximately 20 centers.The expected total study duration is approximately 12-15 months, representing the time necessary to enroll the target sample size and to complete the 3-month follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

Subject will be implanted with a MicraTM (Model MC1AVR1) for an approved indication.

* Subject has history of AV block.
* Subject is ≥ 18 years old and as per required local law.
* Subject (and/or witness as applicable per local regulations) provides signed and dated authorization and/or consent per institution and local requirements.
* Subject is willing and able to comply with the protocol.

Exclusion Criteria:

* Subject currently enrolled or planning to participate in a potentially confounding drug or device trial during the study. Co-enrollment in concurrent trials is only allowed when documented pre-approval is obtained from the Medtronic Clinical Research Specialist.
* Subject implanted with a MicraTM (Model MC1AVR1) on a non-permanent basis (e.g. CIED infection).
* Subject is pregnant (if required by local law, women of child-bearing potential must undergo a pregnancy test within seven days prior to MicraTM Model MC1AVR1 implant procedures).
* Subject meets any exclusion criteria required by local law (age or other).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2020-06-09 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larry Chinitz, MD, Study Chair — NYU Langone
Locations (20):
- United States (18):
  - Saint Joseph's Medical Center, Stockton, California
  - Baptist Medical Center Jacksonville, Jacksonville, Florida
  - Citrus Cardiology Consultants PA, Leesburg, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Catholic Medical Center, Manchester, New Hampshire
  - Northwell Health, Manhasset, New York
  - NYU Langone Medical Center, New York, New York
  - Duke University Nedical Center, Durham, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Mount Carmel Health System, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Centennial Heart Cardiovascular Consultants, Nashville, Tennessee
  - Baylor Research Institute, Plano, Texas
  - Multicare Institute for Research and Innovation, Tacoma, Washington
  - University of Wisconsin (UW) Hospital and Clinics, Madison, Wisconsin
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong, HK
  - Prince of Wales Hospital, Shatin, HK

REFERENCES:
- [Derived] Chinitz LA, El-Chami MF, Sagi V, Garcia H, Hackett FK, Leal M, Whalen P, Henrikson CA, Greenspon AJ, Sheldon T, Stromberg K, Wood N, Fagan DH, Sun Chan JY. Ambulatory atrioventricular synchronous pacing over time using a leadless ventricular pacemaker: Primary results from the AccelAV study. Heart Rhythm. 2023 Jan;20(1):46-54. doi: 10.1016/j.hrthm.2022.08.033. Epub 2022 Sep 6. PMID 36075532

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were considered enrolled at time of informed consent. Subjects were enrolled between 09 June 2020 and 14 September 2021 at 20 study centers in 2 countries.
Pre-assignment Details: Following enrollment, subjects were implanted with the Micra AV device and completed follow-up visits at 1-month and 3-months post implant. The completed cohort includes subjects implanted with the Micra AV device who had a persistent 3rd degree AV block and normal sinus node function at the 1-month visit.
Groups:
- AccelAV Evaluable for Primary Objective: Subjects implanted with the Micra AV device with a 3rd degree AV block and normal sinus node function at 1-month
Period: Overall Study
Arm/Group | AccelAV Evaluable for Primary Objective
Started | 157
Implanted | 152
1-month Visit | 139
Complete Heart Block at 1-month | 56
At Least 500 Evaluable Beats | 54
Completed | 54
Not Completed | 103
Not completed — Death | 1
Not completed — Exited prior to implant | 5
Not completed — Exited prior to 1-month | 9
Not completed — Missed 1-month visit | 3
Not completed — Predominant rhythm exclusion at 1-month | 83
Not completed — Fewer than 500 evaluable beats | 2

BASELINE CHARACTERISTICS:
Groups:
- AccelAV Enrolled Cohort: Subjects enrolled in the AccelAV study
Arm/Group | AccelAV Enrolled Cohort
Number analyzed (Participants) | 157
Age, Categorical [Count of Participants; unit: Participants] — Population: 3 subjects did not have age reported
  Participants
    number analyzed (Participants) | 154
    <=18 years | 0
    Between 18 and 65 years | 17
    >=65 years | 137
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 3 subjects did not have age reported
  years
    number analyzed (Participants) | 154
    (all) | 77.2 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 3 subjects did not have sex reported
  Participants
    number analyzed (Participants) | 154
    Female | 73
    Male | 81
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Hong Kong | 19
  United States | 138
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: BMI was not available for 7 subjects
  kg/m^2
    number analyzed (Participants) | 150
    (all) | 28.2 (7.0)
Comorbidities [Count of Participants; unit: Participants]
  Hypertension | 123
  Atrial fibrillation | 20
  Diabetes | 63
  Coronary Artery Disease | 66
  Myocardial infarction | 12
  Chronic Obstructive Pulmonary Disease | 29
  Dialysis | 13
Preclusion for Transvenous Pacing [Count of Participants; unit: Participants] | 37
Cardiac Perforation Risk [Count of Participants; unit: Participants]
  Low | 74
  Medium | 39
  High | 37
  Unavailable | 7
Pacing Indication [Count of Participants; unit: Participants]
  Bradyarrhythmia with atrial fibrillation (AF) | 5
  Sinus Node Dysfunction | 7
  Atrioventricular (AV) Block | 137
  Syncope | 1
  Other | 4
  Unavailable | 3

OUTCOME MEASURES:

1. Primary Outcome: Atrioventricular (AV) Synchrony During Rest at 1-month Post-implant in Subjects With Persistent 3rd Degree Atrioventrcular Block (AVB) and Normal Sinus Node Function
Description: Atrioventricular synchrony is defined for each P-wave during the 20-minute resting period. Specifically, for each electrocardiogram (ECG) confirmed P-wave that occurs during the 20-minute resting period at the 1-month visit, the endpoint will be considered met if a ventricular beat (ventricular pace or sensed event) is within 300 ms following an ECG confirmed P-wave. The reported percentage is the average percentage of P-waves considered synchronous across all patients during the 20-minute resting period.
Time Frame: 1-month post-implant
Measure: Mean (95% Confidence Interval); unit: Percentage of P-waves
Arm/Group | AccelAV Evaluable for Primary Objective
Number analyzed (Participants) | 54
Percentage of P-waves | 85.4 [81.1 to 88.9]

2. Secondary Outcome: Stability of AV Synchrony During Rest Between 1-month and 3-months Post-implant in Subjects With Persistent 3rd Degree AVB and Normal Sinus Node Function
Description: AV synchrony is defined for each ECG confirmed P-wave that occurs during the 20-minute resting period at both the 1-month visit and 3-months visits. For each P-wave the endpoint will be considered met if a ventricular beat (ventricular pace or sensed event) is within 300 ms following an ECG confirmed P-wave. The reported percentages are the average percentage of P-waves considered synchronous across all patients during the 20-minute resting period at each visit (month 1 or month 3).
Time Frame: Between 1-month and 3-months post-implant
Population: Subjects were required to have a predominant heart rhythm of persistent 3rd degree AV block and normal sinus node function at both the 1-month and 3-month visits. Of the 54 subjects with persistent 3rd degree AV block an normal sinus function at 1-month, 37 of these remained in persistent 3rd degree AV block an normal sinus function at 3-months and were included in the analysis of this objective.
Measure: Mean (95% Confidence Interval); unit: Percentage of P-waves
Groups:
- AccelAV Evaluable for Secondary Objective: Subjects implanted with the Micra AV device with persistent 3rd degree AV block and normal sinus node function at 1-month and 3-months
Arm/Group | AccelAV Evaluable for Secondary Objective
Number analyzed (Participants) | 37
Percentage of P-waves
  AV synchrony at 1-month | 86.1 [81.2 to 89.9]
  AV synchrony at 3-months | 84.1 [78.3 to 88.6]
  Difference in AV Synchrony (Month 3 - Month 1) | -2.0 [-6.8 to 2.9]

3. Secondary Outcome: Percentage of Ambulatory AV Synchrony at 1-month Post-implant in Subjects With Persistent 3rd Degree AVB and Normal Sinus Node Function
Description: AV synchrony is defined for each P-wave during the the 24-hour Holter monitoring period while the subject went about their activities of daily living. Specifically, for each electrocardiogram (ECG) confirmed P-wave that occurs during the 24-hour Holter period at the 1-month visit, the endpoint will be considered met if a ventricular beat (ventricular pace or sensed event) is within 300 ms following an ECG confirmed P-wave. The reported percentage is the average percentage of P-waves considered synchronous across all patients during the 24-hour Holter monitoring period.
Time Frame: 1-month post-implant
Measure: Mean (95% Confidence Interval); unit: Percentage
Arm/Group | AccelAV Evaluable for Primary Objective
Number analyzed (Participants) | 54
Percentage | 74.5 [70.4 to 78.2]

4. Secondary Outcome: Left Ventricular Outflow Tract Velocity Time Integral
Description: Characterize the change in stroke volume, as measured by left ventricular outflow tract (LVOT) velocity time Integral (VTI), during Micra AV mediated VDD (atrioventricular synchronous ventricular pacing) pacing and VVI (asynchronous ventricular pacing) pacing in subjects with persistent 3rd degree AV block and normal sinus node function
Time Frame: Within 48 hours of procedure
Population: The analysis population is a subset of the enrolled population. Specifically, of the 157 enrolled, 78 subjects had a predominant rhythm of persistent 3rd degree AV block and normal sinus rhythm at the time of implant. Of these, 67 had LVOT VTI measurements in both VVI and VDD modes. Of these 67, 47 had a heart rate within 15 beats per minute in both pacing modes and were included in the analysis of this objective as pre-specified in the study protocol.
Measure: Mean (95% Confidence Interval); unit: cm
Groups:
- AccelAV Evaluable for Secondary Objective: Subjects implanted with the Micra AV device with persistent 3rd degree AV block and normal sinus node function at implant with evaluable echocardiogram data.
Arm/Group | AccelAV Evaluable for Secondary Objective
Number analyzed (Participants) | 47
cm
  LVOT VTI during VVI mode | 21.4 [19.7 to 23.1]
  LVOT VTI during VDD mode | 23.7 [21.7 to 25.6]
  LVOT VTI difference (VDD-VVI) | 2.3 [1.5 to 3.1]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of consent through 3-month follow-up
Arm/Group | AccelAV Enrolled Cohort
All-Cause Mortality (participants affected / at risk) | 2/157
Serious Adverse Events (participants affected / at risk) | 45/157
Other Adverse Events (participants affected / at risk) | 27/157
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AccelAV Enrolled Cohort (N=157)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Acute left ventricular failure (Cardiac disorders) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 2 (3)
Atrial fibrillation (Cardiac disorders) | 3 (3)
Atrial flutter (Cardiac disorders) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 4 (4)
Cardiac failure (Cardiac disorders) | 3 (3)
Cardiac failure acute (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 2 (2)
Cardiac tamponade (Cardiac disorders) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Intracardiac thrombus (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 3 (3)
Pericarditis (Cardiac disorders) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (2)
Haemorrhage intracranial (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Device pacing issue (Product Issues) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Aortic stenosis (Vascular disorders) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
Intermittent claudication (Vascular disorders) | 1 (1)
Peripheral vein occlusion (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AccelAV Enrolled Cohort (N=157)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
Implant site erythema (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Oedema (General disorders) | 1 (1)
Pacemaker syndrome (General disorders) | 4 (5)
Puncture site haemorrhage (General disorders) | 1 (1)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Syncope (Nervous system disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
Orthostatic hypotension (Vascular disorders) | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PIs will not publish/present results until a multi-center pub. is released. If a multi-center pub. is not released within 1 year of completion PI may publish the results pertaining to their activities. Pubs will be provided to MDT at least 60 days prior to submission or presentation for review. Within 60 days of receipt, MDT will verify presence of CI or technical errors. PI will make requested changes prior to publication/presentation. PI will delay publication up to 90 more days if requested.

DOCUMENTS (2):
  • Study Protocol (2020-01-24): https://cdn.clinicaltrials.gov/large-docs/45/NCT04245345/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-13): https://cdn.clinicaltrials.gov/large-docs/45/NCT04245345/SAP_001.pdf